CLINICAL TRIAL: NCT02847975
Title: Sodium Nitrate to Improve Blood Flow
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ron Victor, Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00033300
Record Dates: First submitted 2014-04-30; First posted 2016-07-28 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker; dystrophy; sympatholysis
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — sodium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sodium nitrate (Experimental): Sodium nitrate will be administered orally and functional sympatholysis assessed before and after treatment
  Interventions: Dietary Supplement: Sodium nitrate

INTERVENTIONS:
Dietary Supplement: Sodium nitrate — Sodium nitrate will be ingested orally

SUMMARY:
Investigators recently showed that tadalafil restores functional sympatholysis in patients with Becker muscular dystrophy (BMD). If tadalafil restores functional sympatholysis in BMD via the NO-cyclic guanosine monophosphate pathway, then functional sympatholysis should also be restored by sodium nitrite- which is an indirect nitric oxide donor.

ELIGIBILITY:
Inclusion Criteria:

* Becker muscular dystrophy
* age 15-55 years of age
* ambulatory

Exclusion Criteria:

* hypertension, diabetes, or heart failure by standard clinical criteria
* elevated brain natriuretic peptide level (>100 pg/ml)
* Left ventricular ejection fraction < 50%
* cardiac rhythm disorder, specifically: rhythm other than sinus, supraventricular tachycardia, atrial fibrillation, ventricular tachycardia, heart block
* continuous ventilatory support
* liver disease
* renal impairment
* history of asthma or bronchospasm
* use of any medications other than common supplements
* unable to perform handgrip exercise

Ages: 15 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change in muscle tissue oxygenation | change from baseline to post treatment (3-4 hours)
  The pre-specified primary outcome is the pre vs. post treatment change in functional sympatholysis measured by muscle oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
Published http://www.ncbi.nlm.nih.gov/pubmed/26437761

REFERENCES:
- [Background] Martin EA, Barresi R, Byrne BJ, Tsimerinov EI, Scott BL, Walker AE, Gurudevan SV, Anene F, Elashoff RM, Thomas GD, Victor RG. Tadalafil alleviates muscle ischemia in patients with Becker muscular dystrophy. Sci Transl Med. 2012 Nov 28;4(162):162ra155. doi: 10.1126/scitranslmed.3004327. PMID 23197572